CLINICAL TRIAL: NCT03943940
Title: A Preliminary Safety and Efficacy Evaluation of Bone Marrow Mononuclear Cells (BM-MNCs) and Umbilical Cord Tissue-derived Mesenchymal Stem Cells (UC-MSC) Infusion for Type 2 Diabetes Mellitus (T2DM) Patients
Brief Title: BM-MNCs and UC-MSCs Infusion for Type 2 Diabetes Mellitus Patients
Acronym: T2DM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Van Hanh General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNLS012019-TBG
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BM-MNC and UC-MSC (Experimental): 30 patients with Type 2 Diabetes Mellitus will be enrolled and received mononuclear cells and mesenchymal stem cells by intravenous infusion.
  Interventions: Biological: BM-MNC and UC-MSC
- Stand medicines (Other): 30 patients with Type 2 Diabetes Mellitus will be enrolled and treated by standard medicines.
  Interventions: Other: Control

INTERVENTIONS:
Biological: BM-MNC and UC-MSC — Autologous bone marrow mononuclear cells (BM-MNCs) and allogeneic umbilical cord tissue-derived mesenchymal stem cells (UC-MSCs) under sterile conditions to treat this disease.
  UC-MSC: 1-2 x 10^6 cells/kg
  Arms: BM-MNC and UC-MSC
Other: Control — Standard medicine
  Arms: Stand medicines

SUMMARY:
The purpose of this study is to evaluate the preliminary safety and efficacy of autologous bone marrow mononuclear cells (BM-MNCs) and allogeneic umbilical cord tissue-derived mesenchymal stem cells (UC-MSCs) infusion in type 2 Diabetes Mellitus patients.

DETAILED DESCRIPTION:
Mononuclear cells are collected from autologous bone marrow and allogeneic mesenchymal stem cells are isolated and cultured from umbilical cord tissues.

30 patients with Type 2 Diabetes Mellitus will be enrolled and received mononuclear cell and mesenchymal stem cell by intravenous infusion and followed up for 6 months. The other 30 patients with Type 2 Diabetes Mellitus will be enrolled and treated by standard medicines, which would be used as the control group.

Safety is to assess the occurrence of adverse events (AEs) during either stem cells infusion or by physician assessments.

The primary endpoint is to assess the improvement of patient's C-peptid and HOMA-β, HOMA-IR, cytokines TNF-α, IL-1β, Blood glucose level, Hemoglobin A1c (HbA1c) level.

ELIGIBILITY:
Inclusion Criteria:

* Who is diagnosed with Type 2 Diabetes Mellitus according to the ADA 3 years or more
* Patients are able to read, write and understand ICF form and agree to participate in the study
* Males and females between age 18 and 70 years at the screening.
* FBG > 7 mmol/L
* 8% ≤ HbA1C ≤ 11%
* Fasting C-peptide > 0.6 ng/ml
* Anti GAD (-)
* The patient is treated by two oral diabetes medications but uncontrolled blood glucose (HbA1C ≥ 8%)

Exclusion Criteria:

* Pregnant women, planning to become pregnant and lactating women during the study period
* The patient has a disease or a history of vascular disease; history of abdominal or chest aortic disease;
* Patients are diagnosed with heart failure degree IV according to NYHA or kidney failure degree IV according to KDIGO;
* Patients with severe malignancy or dysplasia within 5 years prior to the study period or who are suffering from severe malignant or dysplasia
* Infection is undergoing antibiotic treatment or antibiotics have just been discontinued within 14 days
* Hematologic disease or coagulopathy
* There are abnormalities in liver function (AST and/or ALT ≥ 2 times or bilirubin ≥ 2.0 times normal value at the time of screening);
* Patients with immunodeficiency diseases such as HIV or hepatitis B and C;
* Acute or chronic pancreatitis or a history of acute pancreatitis;
* Patients taking immunosuppressive drugs (such as azathioprine, methotrexate) within 6 months before the study time or taking immunosuppressive drugs;
* The patient is unable to complete the study;
* The patient is participating in another study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
The level of C-peptid and HOMA-β | enrollment, 1 month, 3 months and 6 months after transplantation
  Assess the changes in C-peptid and HOMA-β level after transplantation
The level of HOMA-IR and cytokines TNF-α, IL-1β | enrollment, 1 month, 3 months and 6 months after transplantation
  Assess the changes in HOMA-IR and cytokines TNF-α, IL-1β level after transplantation
Blood glucose level | enrollment, 1 month, 3 months and 6 months after transplantation
  Assess the changes in Blood glucose level after transplantation
Hemoglobin A1c (HbA1c) level | enrollment, 1 month, 3 months and 6 months after transplantation
  Assess the changes in HbA1C level after transplantation
Adverse events | during the course of 6 months
  Number of adverse events in both groups

SECONDARY OUTCOMES:
Insulin dose and drug dosage | enrollment, 1 month, 3 months and 6 months after transplantation
  Assess the changes in Insulin dose and drug dosage after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Thi-Bich Le, MSc-MD, Principal Investigator — Stem Cell Unit, Van Hanh General Hospital
Locations (1):
- Van Hanh General Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam